CLINICAL TRIAL: NCT00003409
Title: A Phase I Dose Escalating Study of the Safety and Tolerability of Gadolinium Texaphyrin as a Radiation Sensitizer in Patients With Primary Glioblastoma Multiforme
Brief Title: Motexafin Gadolinium Plus Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066421; UCLA-HSPC-970904203; COOPER-RP-97-126; LAC-USC-6G971; UCD-RW-98-01; UCLA-HSPC-970904201; UCLA-HSPC-970904202; NCI-T97-0108
Record Dates: First submitted 1999-11-01; First posted 2003-12-02 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — motexafin gadolinium; Radiotherapy

INTERVENTIONS:
Drug: motexafin gadolinium
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Motexafin gadolinium may increase the effectiveness of radiation therapy by making tumor cells more sensitive to radiation.

PURPOSE: Phase I trial to study the effectiveness of motexafin gadolinium plus radiation therapy in treating patients who have newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and tolerability of motexafin gadolinium in combination with radiotherapy in patients with newly diagnosed glioblastoma multiforme. II. Determine the intratumoral pharmacology and quantitative pharmacokinetics of this drug in this patient population.

OUTLINE: This is a multicenter, dose-escalation study of motexafin gadolinium. Patients receive a loading dose regimen comprising motexafin gadolinium IV over 10-15 minutes on days 1-5 or days 1-5 and 8-12 (cohort 7). After the loading dose regimen, patients receive a maintenance regimen comprising motexafin gadolinium IV 3 times weekly for a maximum of 6.5 weeks. Patients also undergo radiotherapy once daily, 5 days a week, for 6.5 weeks. Cohorts of 3-6 patients receive an escalating number of doses of motexafin gadolinium until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Patients are followed at 4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A maximum of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed newly diagnosed glioblastoma multiforme requiring radical radiotherapy No anaplastic astrocytoma or low-grade astrocytoma Able to start radiotherapy within 5 weeks of definitive surgery (unless delay due to cause other than medical illness or poor performance status)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: See Disease Characteristics Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: AST and ALT no greater than 2 times upper limit of normal (ULN) Bilirubin no greater than 2 mg/dL PT and aPTT no greater than 1.5 times ULN Renal: Creatinine less than 1.5 mg/dL Cardiovascular: No severe cardiac disease Pulmonary: No severe lung disease Other: No other significant life-threatening disease No other active malignancy No known glucose-6-phosphate dehydrogenase deficiency No known porphyria Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No biologic therapy for at least 4 weeks after study completion No immunotherapy for at least 4 weeks after study completion Chemotherapy: No chemotherapy for at least 4 weeks after study completion Endocrine therapy: Concurrent steroids allowed Radiotherapy: See Disease Characteristics No prior radiotherapy for this disease or other brain tumor No prior radiotherapy to face, head, or neck Surgery: See Disease Characteristics Recovered from prior surgery or postoperative complication Other: At least 48 hours since prior MRI scan with contrast No concurrent MRI scans with contrast No other concurrent experimental drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-07

CONTACTS AND LOCATIONS:
Overall Officials: Judith M. Ford, MD, PhD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California

REFERENCES:
- [Result] Ford JM, Seiferheld W, Alger JR, Wu G, Endicott TJ, Mehta M, Curran W, Phan SC. Results of the phase I dose-escalating study of motexafin gadolinium with standard radiotherapy in patients with glioblastoma multiforme. Int J Radiat Oncol Biol Phys. 2007 Nov 1;69(3):831-8. doi: 10.1016/j.ijrobp.2007.04.017. Epub 2007 Jun 8. PMID 17560737